CLINICAL TRIAL: NCT02094664
Title: HHOT AIR Study (a Pilot Study): Heated Humidified Oxygen Therapy Compared to Standard Dry Oxygen: An Assessment in Infants With bRonchiolitis
Brief Title: Heated Humidified Oxygen Compared to Dry Oxygen Therapy in Children With Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Responsible Party: Principal Investigator, Diana Chen, Pediatric Pulmonary Fellow, UCSF Benioff Children's Hospital Oakland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-066
Record Dates: First submitted 2014-03-18; First posted 2014-03-24 (Estimated); Results first posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Bronchiolitis; Hypoxemia
Keywords: Heat; Humidification; Oxygen
MeSH Terms: conditions — Bronchiolitis; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard oxygen via nasal cannula (No Intervention): Standard therapy
- Heated and humidified oxygen (Active Comparator): Heated and humified oxygen
  Interventions: Device: Heated and humidified oxygen

INTERVENTIONS:
Device: Heated and humidified oxygen
  Arms: Heated and humidified oxygen

SUMMARY:
The purpose of this study is to compare heat and humidified oxygen with cold and dry oxygen in children with bronchiolitis.

The hypotheses are that heating and humidifying inspired low flow supplemental oxygen will optimize mucociliary function thereby, 1) improve oxygenation, 2) decrease work of breathing, and 3) decrease length of hospital stay.

DETAILED DESCRIPTION:
Bronchiolitis is the leading cause of acute respiratory illness and hospitalization in infants and young children. The mainstay of treatment is supportive care, which includes frequent nasal suctioning, intravenous fluid hydration, and supplemental oxygen for hypoxemia.

The airways normally heat and humidify inspired ambient air to core temperature amd 100% relative humidity at the carina. This environment, at core temperature, allows for optimal mucociliary clearance. Supplemental oxygen delivered via wall source is cold and dry, and does not reach core temperature and 100% humidity until some point distal to the carina, past the main bronchi. This presses on the lower respiratory tract to assist in heat and moisture exchange and thus decrease ciliary function. This, in combination with bronchiolitis, can impair mucociliary clearance.

Specific aim 1: Determine the effect of heated and humidified oxygen therapy on clinical improvement in children with bronchiolitis, based on Respiratory Distress Assessment Instrument (RDAI) and respiratory rate (RR).

Specific aim 2: Determine the effect of heated and humidified oxygen therapy on length of hospital stay and duration of supplemental oxygen requirement in children with bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

* Ages ≤24 months of age
* Physician diagnosed bronchiolitis
* Admitted to pediatric floor
* Supplemental oxygen requirement, <4 L/min, for hypoxemia, oxygen saturation <92% in room air

Exclusion Criteria:

* Prematurity, born <37 weeks gestational age
* Admitted to pediatric intensive care unit for medical indication
* Requirement of heated, humidified high flow system
* Chronic lung disease (such as bronchopulmonary dysplasia, cystic fibrosis, primary ciliary dyskinesia, tracheostomy status, baseline oxygen requirement)
* Neuromuscular disorders
* Chromosomal defects
* Metabolic disorders
* Immunodeficiency
* Unrepaired cardiac abnormalities

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Chen, M.D., Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- Children's Hospital and Research Center Oakland, Oakland, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Standard dry oxygen therapy
- Treatment: Heated and humidified oxygen therapy
Period: Overall Study
Arm/Group | Control | Treatment
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Treatment | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 16 | 32
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 9 | 11 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 1 | 5 | 6
  Ethnicity: Black | 4 | 1 | 5
  Ethnicity: Hispanic | 6 | 6 | 12
  Ethnicity: Other | 5 | 4 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 16 | 32
Mean RDAI [Mean (Standard Deviation); unit: units on a scale] — Respiratory Distress Assessment Instrument (RDAI) is a validated clinical assessment scale used to evaluate severity of respiratory illness in children with bronchiolitis. It is based on 2 variables, wheezing and retractions. Points are applied to each variable to give a score ranging from 0 to 17. Higher total score means subject is clinically more severe.
  units on a scale | 5.38 (3.65) | 4.44 (2.61) | 4.90 (3.16)
Mean RR [Mean (Standard Deviation); unit: bpm] | 45.44 (12.74) | 48.19 (11.3) | 46.8 (11.9)
Mean sick days [Mean (Standard Deviation); unit: days] | 4.56 (1.36) | 4.25 (1.43) | 4.41 (1.39)
Respiratory Syncytial Virus (RSV) positive [Count of Participants; unit: Participants] | 11 | 13 | 24
Family history of asthma [Count of Participants; unit: Participants] | 6 | 8 | 14
Smoke exposure at home [Count of Participants; unit: Participants] | 6 | 3 | 9
Inhaled albuterol in emergency department [Count of Participants; unit: Participants] | 10 | 9 | 19
Systemic steroids in emergency department [Count of Participants; unit: Participants] | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Respiratory Distress Assessment Instrument (RDAI) From Baseline.
Description: The RDAI is a validated clinical scoring system to assess respiratory distress and has been used in several bronchiolitis studies. The RDAI is based on two variables, wheezing and retractions, in which points are applied to each to give a score ranging from 0 to 17. The higher the total score, the worse the subject was clinically. Reported are the absolute scores at each time point, for each arm. Baseline scores are reported in the Baseline Module.
Time Frame: Baseline, Hour 1, Hour 4, Hour 8, and Hour 12
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control: Standard dry therapy therapy
Arm/Group | Control | Treatment
Number analyzed (Participants) | 16 | 16
units on a scale
  Hour 1 | 4.69 (3.4) | 2.69 (3.2)
  Hour 4 | 4.27 (3.01) | 3 (2.63)
  Hour 8 | 4.33 (3.34) | 3.44 (3.2)
  Hour 12 | 3.64 (2.25) | 3.2 (2.37)

2. Primary Outcome: Change in Respiratory Rate (RR) From Baseline
Description: Respiratory rate was measured by counting respirations for one minute. Reported are the absolute scores at each time point, for each arm. Baseline scores are reported in the Baseline Module.
Time Frame: Baseline, Hour 1, Hour 4, Hour 8, and Hour 12
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Control | Treatment
Number analyzed (Participants) | 16 | 16
breaths per minute
  Baseline | 45.44 (12.74) | 48.19 (11.3)
  Hour 1 | 44.81 (12.69) | 45.81 (12.16)
  Hour 4 | 45.73 (14.26) | 47.25 (8.84)
  Hour 8 | 43.75 (8.06) | 43.44 (8.74)
  Hour 12 | 43.36 (8.54) | 44.93 (9.92)

3. Secondary Outcome: Length of Hospital Stay
Description: Length of hospital stay is measured in days and counted from day of admission to day of discharge.
Time Frame: Subjects will be followed for the duration of hospital stay until discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control | Treatment
Number analyzed (Participants) | 16 | 16
days | 4.44 (2.31) | 4.56 (4.1)

4. Secondary Outcome: Duration of O2 Use
Description: Duration on supplemental O2 was measured in hours.
Time Frame: Subjects will be followed for the duration of oxygen requirement until oxygen discontinued
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Control | Treatment
Number analyzed (Participants) | 16 | 16
hours | 60.02 (48.93) | 72.11 (75.38)

ADVERSE EVENTS:
Arm/Group | Control | Treatment
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No